CLINICAL TRIAL: NCT04550650
Title: Follow-up Study of the Effectiveness of Virtual Reality Therapy in MS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Dr. József Tollár, Head of Neurorehabilitation ,7400 Kaposvár, Tallián Gy. u 20-32, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB2020/08
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Primary Progressive
Keywords: multiple sclerosis; posture; neurorehabilitation; balance
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Controll (No Intervention): No intervention
- Training grp (Experimental): Neurorehabilitation 2 years long intervention, administered daily, targeted postural instability, balance and mobility using at-limit intensity sensorimotor and visuomotor agility training
  Interventions: Other: Training groupe
- PNF (Experimental): 2 years long, You have only treated patients with the PNF technique.
  Interventions: Other: PNF
- Spinning group (Experimental): Patients developed endurance for 2 years. They worked using a spinning bike.
  Interventions: Other: Spinning grp
- Balance (Experimental): Neurorehabilitation 2 years long intervention, administered daily, targeted postural instability, balance
  Interventions: Other: Balance

INTERVENTIONS:
Other: Training groupe — Using virtual training
  Arms: Training grp
Other: PNF — PNF technique was used
  Arms: PNF
Other: Spinning grp — They only worked with spinning bikes.
  Arms: Spinning group
Other: Balance — Balance development was done
  Arms: Balance

SUMMARY:
Different therapies can improve clinical and motor symptoms of multiple sclerosis (MS) similarly, but studies comparing the effects of different exercise therapies on clinical and motor outcomes are scant. We compared the effects of exergaming (EXE), balance (BAL), cycling (CYC), proprioceptive neuromuscular facilitation (PNF), and a standard care wait-listed control group (CON) on clinical and motor symptoms and quality of life (QoL) in people with MS (PwMS).

Methods: PwMS (n = 68, 90% female; age, 47.0 yr; Expanded Disability Status Scale score 5-6) were randomized into five groups. Before and after the interventions (five times a week for 5 wk), PwMS were tested for MS-related clinical and motor symptoms (Multiple Sclerosis Impact Scale-29 (MSIS-29), primary outcome), QoL (EuroQol Five Dimensions Questionnaire), symptoms of depression, gait and balance ability (Tinetti Assessment Tool), static and dynamic balance and fall risk (Berg Balance Scale), walking capacity (6-min walk test), and standing posturography on a force platform.

Patients were followed up for 2 years after 5 weeks of intensive care. Tests are performed every six months.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis
* instability problem

Exclusion Criteria:

• Severe heart problems, severe demeanor, alcoholism, drug problems

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Postural instability | 2 years
  Body sway (mm) (Posturography test)
EQ-5D quality of life | 2 years
  EQ-5D (EQ-5D was first introduced in 1990 by the EuroQol Group, The EQ-5D questionnaire is made up for two components; health state description and evaluation)
balance test | 2 years
  Berg Balance test (The Berg Balance Scale (BBS) was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks, 41-56 = low fall risk, 21-40 = medium fall risk, 0 -20 = high fall risk )
mobility test | 2 years
  Six minutes walk test (6MWT) (m) (The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway)
depression scale | 2 years
  Beck Depression scale (The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression, 0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, 29-63: severe depression)
MSIS-29 | 2 years
  Multiple Sclerosis Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=MS+rehabilitation